CLINICAL TRIAL: NCT01630967
Title: A Phase II Single Arm Study of Degarelix in Men With Castrate Resistant Prostate Cancer With a Rising Prostate-Specific Antigen (PSA) Despite LHRH Agonist Therapy.
Brief Title: Efficacy Study of Switching to a Lutenizing Hormone-releasing Hormone (LHRH) Antagonist From a LHRH Agonist to Treat Progressive Castrate Resistant Prostate Cancer (CRPC)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: British Columbia Cancer Agency (Other)
Collaborators: Ferring Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Kim Chi, Associate Professor of Medicine, University of British Columbia, British Columbia Cancer Agency
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BCCA_Deg01
Record Dates: First submitted 2012-06-25; First posted 2012-06-28 (Estimated); Last update posted 2012-06-28 (Estimated); Status verified 2012-06

CONDITIONS: Prostate Neoplasm
Keywords: castrate resistance; PSA progression; LHRH antagonism
MeSH Terms: conditions — Prostatic Neoplasms | interventions — acetyl-2-naphthylalanyl-3-chlorophenylalanyl-1-oxohexadecyl-seryl-4-aminophenylalanyl(hydroorotyl)-4-aminophenylalanyl(carbamoyl)-leucyl-ILys-prolyl-alaninamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Degarelix (Experimental): Degarelix 240mg subcutaneously loading dose, then 80mg sc every month until disease progression.
  Interventions: Drug: Degarelix

INTERVENTIONS:
Drug: Degarelix — Standard dosing and schedule for administration of degarelix will be used. 240mg s.c. loading dose, 80mg s.c. monthly maintenance dose.
  Other Names: Firmagon

SUMMARY:
Men with castrate resistant prostate cancer who are switched from a luteinizing hormone-releasing hormone (LHRH) antagonists from a LHRH agonist will experience a fall in prostate-specific antigen (PSA).

DETAILED DESCRIPTION:
To determine the proportion of patients with castrate resistant Prostate Cancer who have a PSA decline of ≥50% from baseline PSA when switched from an LHRH agonist to an LHRH antagonist.

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed adenocarcinoma of the prostate
* currently receiving LHRH agonist
* Anti-androgen oral therapy is permitted but will be discontinued upon enrollment
* PSA > 2 ng/ml
* rising PSA despite LHRH agonist
* patients may or may not have clinical evidence off metastases. If metastases are present, they must be asymptomatic and in bone or lymph node only
* Prior chemotherapy allowed
* ECOG performance status 0-1

Exclusion Criteria:

* Patients with a history of other active malignancies, except: adequately treated non-melanoma skin cancer, superficial bladder cancer, or other solid tumours curatively treated with no evidence of disease for ≥ 3 years.
* Other serious illness, psychiatric or medical condition that would not permit the patient to be managed according to the protocol including: i)Significant cardiovascular condition including but not limited to: uncontrolled hypertension, unstable angina, significant congestive heart failure or myocardial infarction, deep venous thrombosis, pulmonary embolus or cerebrovascular attack within the last 6 months. ii) History of significant neurological disorder that would impair the ability to obtain consent

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2012-08; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
50% fall in PSA | 8 weekly
  Proportion of patients with castrate resistant prostate cancer (CRPC) who have a PSA decline of ≥50% from baseline when switched from an LHRH agonist to an LHRH antagonist

SECONDARY OUTCOMES:
Luteinizing hormone (LH) | 8 weekly
  Circulating androgen and pituitary hormones will be measured during the course of the study (8 weekly).
Follicle stimulating hormone (FSH) | 8 weekly
  Circulating androgen and pituitary hormones will be measured during the course of the study (8 weekly).
Testosterone (TT) | 8 weekly
  Circulating androgen and pituitary hormones will be measured during the course of the study (8 weekly).
dehydroepiandrosterone (DHEA) | 8 weekly
  Circulating androgen and pituitary hormones will be measured during the course of the study (8 weekly).
dehydroepiandrosterone-sulfate (DHEA-S) | 8 weekly
  Circulating androgen and pituitary hormones will be measured during the course of the study (8 weekly).
androstenedione (AED) | 8 weekly
  Circulating androgen and pituitary hormones will be measured during the course of the study (8 weekly).
dihydrotestosterone (DHT) | 8 weekly
  Circulating androgen and pituitary hormones will be measured during the course of the study (8 weekly).

CONTACTS AND LOCATIONS:
Overall Officials: Kim N Chi, MD, Principal Investigator — British Columbia Cancer Agency, Univeristy of British Columbia
Locations (1):
- British Columbia Cancer Agency, Vancouver, British Columbia, Canada

REFERENCES:
- [Result] Crawford ED, Tombal B, Miller K, Boccon-Gibod L, Schroder F, Shore N, Moul JW, Jensen JK, Olesen TK, Persson BE. A phase III extension trial with a 1-arm crossover from leuprolide to degarelix: comparison of gonadotropin-releasing hormone agonist and antagonist effect on prostate cancer. J Urol. 2011 Sep;186(3):889-97. doi: 10.1016/j.juro.2011.04.083. Epub 2011 Jul 23. PMID 21788033